CLINICAL TRIAL: NCT01221532
Title: Support From Hospital to Home for Elders: A Randomized Controlled Study
Acronym: SHHE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Gordon and Betty Moore Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SHHE2010
Record Dates: First submitted 2010-07-13; First posted 2010-10-15 (Estimated); Last update posted 2013-07-09 (Estimated); Status verified 2013-07

CONDITIONS: Hospital Readmissions

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- SHHE Peridischarge intervention (Experimental): Patients receive the Support from Hospital to Home (SHHE) Peridischarge Intervention plus usual care
  Interventions: Behavioral: SHHE Peridischarge Intervention
- Usual Care (No Intervention)

INTERVENTIONS:
Behavioral: SHHE Peridischarge Intervention — Support from Hospital to Home (SHHE) Peridischarge Intervention patients will receive Usual care plus
  1. a visit with in-hospital registered nurse, who provides additional patient education, assesses patient's needs post-hospitalization, communicates with the medical team, and develops a personalized discharge plan;
  2. two phone calls from a nurse practitioner(NP)/physician assistant (PA) after discharge, in which adherence to medications, treatment plan, and access to outpatient care, and other issues identified during the hospitalization will be explored;
  3. the provision of a phone support line, on which an NP/PA will call patients back within 24 hours to answer questions and assist transition to outpatient care.
  Arms: SHHE Peridischarge intervention

SUMMARY:
The investigators will randomize 700 non-psychiatric, non-obstetric, non-surgical patients aged 55 years and older at San Francisco General Hospital (SFGH) to usual care (ten days of prescription medication, discharge summary sent to primary care provider (PCP), and outpatient appt made for patient, and patient's nurse reviews discharge plan,) or usual care plus a peridischarge intervention (a visit with specialized in-hospital discharge nurse, development of personalized discharge plan, two phone calls from a nurse practitioner(NP)/physician assistant (PA) after discharge and availability of additional calls back from NP/PA, upon patient request, to help answer questions and assist patient's transition to outpatient care, and communication with primary care/subspecialty providers). The usual care and usual care plus intervention groups will be assessed for differences in mortality and rates of rehospitalization and emergency department use 30, 90 and 180 days following discharge from the hospital.

The discharge process from the hospital to home is frequently marked by poor quality and high risk of adverse events and readmissions. It has been hypothesized that better coordinated care, personalized patient education, and follow-up calls to identify potential sources of adverse events, such as medical complications and medication errors can reduce rehospitalization and emergency room visits following discharge from the hospital. Although these interventions have been shown to reduce combined hospital readmissions and emergency department visits in English-speaking patients, none has focused on elderly patients in a diverse urban public hospital setting that includes non-English-speakers, who might benefit more than other populations from enhanced services during and after discharge from the hospital. Further, these labor-intensive interventions are costly to implement, and it is unknown whether opportunity cost of providing additional services in a limited-resource environment such as San Francisco General Hospital (SFGH) outweighs the unknown clinical benefits.

ELIGIBILITY:
Inclusion Criteria:

* patients age 55 and older
* admitted to the general medicine, family medicine, cardiology, and neurology services at San Francisco General Hospital,
* able to communicate in either English, Spanish, Mandarin or Cantonese,
* attending physicians agree to the patient's participation.
* Patients must be able to demonstrate an understanding of the study's goals through a set of teach back questions included in the consent process.

Exclusion Criteria:

* transferred from an outside hospital;
* admitted for a planned hospitalization (e.g. chemotherapy, a planned surgery)
* requiring hospice, nursing home, rehab or other institutional settings (i.e. expected by the physician team to be discharged to skilled nursing facilities) - those unable to independently consent (i.e. severely cognitively impaired, delirious, deaf, or involuntarily hospitalized because of severe mental illness)
* unable to understand English, Spanish or Cantonese (as reported by medical teams or unable to complete the consent teach-back process)
* less than age 55
* aphasic
* otherwise excluded by the medical team
* participated in the pilot project of this intervention.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 699 (Actual)
Dates: Start 2010-07; Primary Completion 2012-02 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Combined Emergency Department Visits and Inpatient Readmissions | 30 days after discharge from hospital
Combined Emergency Department Visits and Inpatient Readmissions | 90 days after discharge from hospital
Combined Emergency Department Visits and Inpatient Readmissions | 180 days after discharge from hospital

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey M Critchfield, MD, Principal Investigator — University of California, San Francisco; Sue Currin, RN, Principal Investigator — San Francisco General Hospital
Locations (1):
- San Francisco General Hospital, San Francisco, California, United States

REFERENCES:
- [Derived] Chan B, Goldman LE, Sarkar U, Guzman D, Critchfield J, Saha S, Kushel M. High perceived social support and hospital readmissions in an older multi-ethnic, limited English proficiency, safety-net population. BMC Health Serv Res. 2019 May 24;19(1):334. doi: 10.1186/s12913-019-4162-6. PMID 31126336
- [Derived] Chan B, Goldman LE, Sarkar U, Schneidermann M, Kessell E, Guzman D, Critchfield J, Kushel M. The Effect of a Care Transition Intervention on the Patient Experience of Older Multi-Lingual Adults in the Safety Net: Results of a Randomized Controlled Trial. J Gen Intern Med. 2015 Dec;30(12):1788-94. doi: 10.1007/s11606-015-3362-y. PMID 25986136
- [Derived] Goldman LE, Sarkar U, Kessell E, Guzman D, Schneidermann M, Pierluissi E, Walter B, Vittinghoff E, Critchfield J, Kushel M. Support from hospital to home for elders: a randomized trial. Ann Intern Med. 2014 Oct 7;161(7):472-81. doi: 10.7326/M14-0094. PMID 25285540